CLINICAL TRIAL: NCT01264718
Title: A Randomized Trial of Effects of Parent Mentors on Insuring Minority Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Glenn Flores, MD, Professor, Chief Research Officer, and Associate Chair of Research, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 082010-138
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Uninsured Children Eligible for Medicaid or CHIP
Keywords: minority health; child; Medicaid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): After randomization to the control group, minority low-income parents of uninsured, Medicaid/CHIP-eligible children received only traditional Medicaid/Children's Health Insurance Program (CHIP) outreach and enrollment.
- Parent Mentors (Experimental): After randomization to the Parent Mentor group, minority low-income parents of uninsured Medicaid/CHIP-eligible children received face-to-face instruction and guidance from Parent Mentors on obtaining and keeping Medicaid/CHIP for their child; getting a doctor, dentist, and pharmacist; and addressing social determinants of health.
  Interventions: Behavioral: Parent Mentors

INTERVENTIONS:
Behavioral: Parent Mentors — After random assignment to the Parent Mentor group, minority low-income parents of Medicaid/CHIP eligible children met with Parent Mentors to receive instruction and help on completing, submitting applications for, and maintaining Medicaid/CHIP coverage for their child.
  Other Names: Kids' HELP
  Arms: Parent Mentors

SUMMARY:
The Kids' HELP trial rigorously documented that a Parent Mentor intervention results in multiple benefits: more children are insured faster, children's access to healthcare and parental satisfaction improve, quality of well-child care is enhanced, thousands of dollars are saved per child, jobs are created, disparities are eliminated, and the intervention potentially could save our nation billions of dollars.

DETAILED DESCRIPTION:
Background: Six million US children are uninsured, despite two-thirds being eligible for Medicaid/Children's Health Insurance Program (CHIP), and minority children are at especially high risk. The most effective way to insure uninsured children, however, is unclear.

Methods: We conducted a randomized trial of the effects of parent mentors (PMs) on insuring uninsured minority children. PMs were experienced parents with >=1 Medicaid/CHIP-covered child who received 2 days of training, then assisted families for 1 year with insurance applications, retaining coverage, medical homes, and social needs; controls received traditional Medicaid/CHIP outreach. The primary outcome was obtaining insurance 1 year post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. The parent/guardian is a primary caretaker of a least one child 0-18 years old who currently has no health insurance
2. The parent/guardian self-identifies the uninsured child as Hispanic/Latino, African-American/Black, or both
3. The uninsured child is eligible for either Medicaid or CHIP
4. The parent/guardian is willing to be contacted monthly by telephone, or in the form of a home visit (if no functioning telephone is present in the household).

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 329 (Actual)
Dates: Start 2010-12; Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Flores, M.D., Principal Investigator — Connecticut Children's Medical Center
Locations (2):
- United States (2):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flores G, Walker C, Lin H, Lee M, Fierro M, Henry M, Massey K, Portillo A. Design, methods, and baseline characteristics of the Kids' Health Insurance by Educating Lots of Parents (Kids' HELP) trial: a randomized, controlled trial of the effectiveness of parent mentors in insuring uninsured minority children. Contemp Clin Trials. 2015 Jan;40:124-37. doi: 10.1016/j.cct.2014.11.015. Epub 2014 Dec 2. PMID 25476583
- [Background] Flores G, Walker C, Lin H, Lee M, Fierro M, Henry M, Massey K, Portillo A. A successful program for training parent mentors to provide assistance with obtaining health insurance for uninsured children. Acad Pediatr. 2015 May-Jun;15(3):275-81. doi: 10.1016/j.acap.2014.09.011. Epub 2014 Dec 1. PMID 25447369
- [Background] Flores G, Lin H, Walker C, Lee M, Currie JM, Allgeyer R, Fierro M, Henry M, Portillo A, Massey K. Parent Mentors and Insuring Uninsured Children: A Randomized Controlled Trial. Pediatrics. 2016 Apr;137(4):e20153519. doi: 10.1542/peds.2015-3519. Epub 2016 Mar 17. PMID 27244706
- [Background] Flores G, Lin H, Walker C, Lee M, Portillo A, Henry M, Fierro M, Massey K. A cross-sectional study of parental awareness of and reasons for lack of health insurance among minority children, and the impact on health, access to care, and unmet needs. Int J Equity Health. 2016 Mar 22;15:44. doi: 10.1186/s12939-016-0331-y. PMID 27000795
- [Background] Flores G, Portillo A, Lin H, Walker C, Fierro M, Henry M, Massey K. A successful approach to minimizing attrition in racial/ethnic minority, low-income populations. Contemp Clin Trials Commun. 2017 Mar;5:168-174. doi: 10.1016/j.conctc.2017.01.009. Epub 2017 Feb 14. PMID 28378019
- See also: Manuscript: Design, methods, and baseline characteristics of the Kids' Health Insurance by Educating Lots of Parents (Kids' HELP) trial: A randomized, controlled trial of the effectiveness of parent mentors in insuring uninsured minority children — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4314321/
- See also: Manuscript: A successful program for training parent mentors to provide assistance with obtaining health insurance for uninsured children — https://www.ncbi.nlm.nih.gov/pubmed/?term=A+successful+program+for+training+parent+mentors+to+provide+assistance+with+obtaining+health+insurance+for+uninsured+children
- See also: Manuscript: A cross-sectional study of parental awareness of and reasons for lack of health insurance among minority children, and the impact on health, access to care, and unmet needs — http://equityhealthj.biomedcentral.com/articles/10.1186/s12939-016-0331-y

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Parent Mentors: Families assisted for one year with insurance applications, retaining coverage, medical homes, and social needs by experienced parents (Parent Mentors) with at least one Medicaid/CHIP-covered child who received two days of training.
- Control: No Intervention: Families received traditional Medicaid/CHIP outreach
Period: Overall Study
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
Started | 172 | 157
Completed | 123 | 114
Not Completed | 49 | 43
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 9 | 15
Not completed — Loss of Medicaid/CHIP eligibility | 37 | 26

BASELINE CHARACTERISTICS:
Population: 237 included in primary analysis: 123 from the intervention group (37 excluded due to loss of Medicaid/CHIP eligibility, 3 were lost to follow-up, and 9 withdrew prior to one-year follow-up); and 114 from the control group (26 due to loss of Medicaid/CHIP eligibility, 2 were lost to follow-up, and 15 withdrew prior to one-year follow-up)
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Parent Mentors | Control: No Intervention | Total
Number analyzed (Participants) | 123 | 114 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 123 | 114 | 237
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7 [3 to 10] | 7 [4 to 12] | 7 [3 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 47 | 119
  Male | 51 | 67 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino | 80 | 75 | 155
  African-American/Black | 43 | 39 | 82
Region of Enrollment [Number; unit: participants]
  United States | 123 | 114 | 237
Number of months child had been uninsured [Median (Inter-Quartile Range); unit: participants] | 6 [4 to 12] | 8 [3 to 24] | 7 [3 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Number of Children With Health Insurance
Description: A study child is considered insured once official written notification of insurance is confirmed, either through an electronic or hard copy of the state coverage letter, or via verification from the Texas Health and Human Services Center.
Time Frame: One year after enrollment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
Number analyzed (Participants) | 123 | 114
Participants
  Child obtained health insurance | 117 | 78
  Child did not obtain health insurance | 6 | 36

2. Secondary Outcome: Number of Days From Study Enrollment to Obtaining Coverage
Description: Zero time (the point at which the maneuver is imposed) is the data and time of study enrollment. Occurrence of the main outcome event is the date and time of official notification that the child is insured.
Time Frame: One year after enrollment
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
Number analyzed (Participants) | 123 | 114
Days | 62 [33 to 112] | 140 [61 to 236]

3. Secondary Outcome: Parental Satisfaction With the Process of Obtaining Coverage for Child
Description: Parental satisfaction is assessed both using a five-point Likert-scale and open-ended questions
Time Frame: One year after enrollment
Population: 121 from the intervention group (37 excluded due to loss of Medicaid/CHIP eligibility, 3 were lost to follow-up, 9 withdrew prior to one-year follow-up, 2 did not answer); and 113 from the control group (26 due to loss of Medicaid/CHIP eligibility, 2 were lost to follow-up, 15 withdrew prior to one-year follow-up, and 1 did not answer).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
Number analyzed (Participants) | 121 | 113
Participants
  1- Parent very unsatisfied with process | 2 | 13
  2- Parent unsatisfied with process | 5 | 10
  3- Parent uncertain about process | 12 | 17
  4- Parent satisfied with process | 33 | 45
  5- Parent very satisfied with process | 69 | 28

4. Secondary Outcome: Intervention Cost-Effectiveness Ratio (ICER)
Description: The difference in total costs between the intervention group and controls
Time Frame: One year after enrollment
Population: as for baseline characteristics
Measure: Number; unit: Dollars
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
Number analyzed (Participants) | 123 | 114
Dollars
  PM stipends- total cost | 53,838 | 0
  PM travel and supplies- total cost | 5,195 | 0
  PM training sessions and meetings- total cost | 1411.61 | 0
  Program coordinator salary- total cost | 25,350 | 0
  ED visits- total cost | 60,885 | 62,730
  Hospitalizations- total cost | 58,431 | 81,537
  ICU stays- total cost | 74,742 | 277,094
  Wage loss/other costs of caring for sick child | 12,985 | 33,589
  Total for all costs | 291,426 | 454,647
Statistical Analysis 1: Comparison: Intervention: Parent Mentors; Test type: Other — The Intervention Cost-Effectiveness Ratio (ICER) is the difference in total costs between the intervention group and controls was divided by the intergroup difference in the proportion of insured children; ICER = 6,045.22 — The estimated value is the savings per child per year insured
Statistical Analysis 2: Comparison: Intervention: Parent Mentors; Test type: Other — [test comment as in outcome 4, analysis 1]; ICER = 4,185.15 — The estimated value is the savings for each percent increase in children obtaining insurance per year

ADVERSE EVENTS:
Time Frame: This project involved a behavioral intervention (not a drug- or device-based intervention), so no participants were at risk of adverse events and no adverse event assessment process was instituted.
Description: This project involved a behavioral intervention (not a drug- or device-based intervention), so no participants were at risk of adverse events and no adverse event assessment process was instituted.
Arm/Group | Intervention: Parent Mentors | Control: No Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No